CLINICAL TRIAL: NCT02952430
Title: Emergency Laparotomy and Frailty; a National Multicentre Prospective Cohort Study of Older Surgical Patients (ELF Study)
Brief Title: Emergency Laparotomy and Frailty Study
Acronym: ELF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: North Western Research Collaborative (Network)
Collaborators: Older persons Surgical Outcomes Collaboration (Unknown)
Responsible Party: Sponsor
Other Study IDs: NWRC- ELF
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Emergencies; Frail Older Adult; Laparotomy
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Frail: Patients over 65 year old having emergency laparotomy with a Frailty score (Modified Rockwood score) of greater than or equal to five.
  This group will then be observed after intervention to review outcomes.
  Interventions: Procedure: Emergency laparotomy
- Not frail: Patients over 65 year old having emergency laparotomy with a Frailty score (Modified Rockwood score) of less than five.
  This group will then be observed after intervention to review outcomes.
  Interventions: Procedure: Emergency laparotomy

INTERVENTIONS:
Procedure: Emergency laparotomy — Patients already undergoing emergency laparotomy - groups divided pre-operatively into frail and not frail based on modified Rockwood score. Then outcomes observed.

SUMMARY:
Patients aged over 65 comprise more than half the emergency general surgical workload, however, available risk-prediction tools for such patients are extrapolated from younger cohorts. Research suggests that high pre-operative frailty scores correlate with increased post-operative mortality and morbidity. Validated frailty assessments may help identify high risk older emergency surgical patients, facilitating decision-making and informing patient choice.

We propose the first prospective UK observational study assessing frailty as an independent predictor of outcome in the older surgical patient undergoing emergency laparotomy.

Prospective data collection of patients over 65 undergoing emergency laparotomy will be performed in 20 NHS Trusts. Pre-operative frailty scores will be evaluated using the Rockwood Frailty Scale. Primary outcome measure is 30-day mortality. Secondary outcome measures are post-operative complications, altered independence status and length of stay.

Results will be disseminated at national/international surgical meetings and published in a peer-reviewed journal.

DETAILED DESCRIPTION:
The ELF steering committee will run this project as part of the North West Research Collaborative(NWRC), consisting of surgical trainees with a successful record of publishing credible research and establishing clinical trials.

Following ethical approval, data will be collected from NHS Trusts throughout the UK. Trained leads will facilitate data collection adhering to a study protocol and local clinical governance.

Patients over 65 undergoing emergency laparotomy will be identified prospectively over 3 months. Demographics, time to surgical intervention, length of stay(LOS), pre- and post-admission independence, intermediate care stay, Clavien-Dindo post-operative complications, 30-day mortality and 30-day re-admission data will be collected on a secure database. Pre-operative frailty will be assessed using the Rockwood Frailty Scale.

500 patients are required for a statistically significant difference in primary outcome (30 day mortality). Secondary outcome measures are complications, change in independence status and LOS. Outcomes will be analysed to compare the impact of frailty.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older
* Admitted to emergency surgical departments
* Requiring an emergency laparotomy

Exclusion Criteria:

- Patients less than 65 years old

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the emergency surgical department requiring an emergency laparotomy
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Mortality | 90 days
  Patient alive at 90 days (rounded up to the nearest whole day) post operatively

SECONDARY OUTCOMES:
Post-operative complications | 30 days
  Evidence of post-operative complications at 30 days (rounded up to the nearest whole day) post operatively. Measured using the Clavein Dindo classification
Lowering of independence status post-operatively | 30 days
  Change in living status from pre to post operatively. Including increased care required at home and discharge to increased care (such as residential or nursing home care).
Length of stay | 30 days
  Length of hospital admission - rounded up to whole days
Readmission | 30 days
  All cause readmission to hospital for emergency care - within 30 days post-operatively (rounded up to the nearest whole day).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Moug, MBChB, PhD, Principal Investigator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bisset CN, Carter B, Law J, Hewitt J, Parmar K, Moug SJ; ELF Study Group Collaborative Authorship. The influence of social media on recruitment to surgical trials. BMC Med Res Methodol. 2020 Jul 28;20(1):201. doi: 10.1186/s12874-020-01072-1. PMID 32723388
- [Derived] Parmar KL, Law J, Carter B, Hewitt J, Boyle JM, Casey P, Maitra I, Farrell IS, Pearce L, Moug SJ; ELF Study Group. Frailty in Older Patients Undergoing Emergency Laparotomy: Results From the UK Observational Emergency Laparotomy and Frailty (ELF) Study. Ann Surg. 2021 Apr 1;273(4):709-718. doi: 10.1097/SLA.0000000000003402. PMID 31188201
- [Derived] Parmar KL, Pearce L, Farrell I, Hewitt J, Moug S. Influence of frailty in older patients undergoing emergency laparotomy: a UK-based observational study. BMJ Open. 2017 Oct 6;7(10):e017928. doi: 10.1136/bmjopen-2017-017928. PMID 28988184